CLINICAL TRIAL: NCT03359135
Title: Compression Garments Effects on Postural Balance of Patients With Hypermobility Type of Ehlers-danlos Syndrome, a Prospective Study on 40 Patients
Brief Title: Compression Garments on Hypermobility Type of Ehlers-Danlos Syndrome (CGhEDS)
Acronym: VECO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hôpital Raymond Poincaré (Other)
Responsible Party: Sponsor
Other Study IDs: hEDS-40
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Hypermobility Type Ehlers-Danlos Syndrome
Keywords: Compression garment
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3 | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group1: hEDS treated with rehabilitation only
  Interventions: Other: Rehabilitation
- group 2: hEDS treated with rehabilitation associated to compression garments wearing
  Interventions: Other: Rehabilitation; Device: Compression Garment

INTERVENTIONS:
Other: Rehabilitation — Rehabilitation during 4 weeks
Device: Compression Garment — Rehabilitation associated to wearing CG during 4 weeks
  Groups: group 2

SUMMARY:
This study evaluates the effects of wearing a compression garment on the postural balance of patients with hypermobility type of Ehlers-Danlos syndrome, in randomised controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years
* hEDS with the 2017 diagnostic criteria .
* A normal neurological examination with no sensory disorders, no cerebellar syndrome or vestibular syndrome.
* An optimal balanced analgesic treatment before inclusion
* Patients who have not modified their physical treatment (physiotherapy) since 6 months.

Exclusion Criteria:

* Surgery of the lower limb (hip, knee or ankle)
* Patient having already wear compression garments in the year preceding.
* Neurological history of sensory , vestibular or cerebellar disorders.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hypermobility type of Ehlers-Danlos syndrome
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Centre of pression speed | 4 weeks
  a stability parameter on a force plate

CONTACTS AND LOCATIONS:
Locations (1):
- Gader Nadra, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benistan K, Foy M, Gillas F, Genet F, Kane M, Barbot F, Vaugier I, Bonnyaud C, Gader N. Effects of compression garments on balance in hypermobile Ehlers-Danlos syndrome: a randomized controlled trial. Disabil Rehabil. 2024 May;46(9):1841-1850. doi: 10.1080/09638288.2023.2209742. Epub 2023 May 17. PMID 37194618